CLINICAL TRIAL: NCT01507857
Title: A Multicentered, Double - Blind, Randomized, and Placebo - Controlled Clinical Trial With Inactivated Enterovirus Type 71 (EV71) Vaccines
Brief Title: An Efficacy Trial in Inactivated Enterovirus Type 71 (EV71) Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-EV71-3001
Record Dates: First submitted 2012-01-02; First posted 2012-01-11 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-03

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: EV71 vaccine; HFMD; efficacy; EV71 associated disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 400U /0.5ml in infants (Experimental): inactivated vaccine(vero cell) against EV71 of 400U /0.5ml in 5000 infants aged 6-35 months old on day0,28
  Interventions: Biological: 400U /0.5ml EV71 vaccine
- 0/0.5ml placebo in infants (Placebo Comparator): 0/0.5ml placebo in 5000 infants aged 6-35 months old on day0,28
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: 400U /0.5ml EV71 vaccine — inactivated vaccine (vero cell) against EV71 of 400U /0.5ml, two doses, 28 days interval
  Other Names: EV71 vaccine
  Arms: 400U /0.5ml in infants
Biological: 0/0.5ml placebo — 0/0.5ml placebo, two doses, 28 days interval
  Other Names: placebo
  Arms: 0/0.5ml placebo in infants

SUMMARY:
The purpose of this study is to evaluate the efficacy, immunogenicity and safety of EV71 Vaccines in preventing Hand, Foot and Mouth disease caused by EV71 in a total 10,000 healthy infants volunteers aged from 6 to 35months old.

DETAILED DESCRIPTION:
The phase II study of inactivated vaccine (vero cell) against EV71 has completed on Dec 2011 in China. The data from the phase I and II study suggested that the inactivated EV71 vaccine had a clinically acceptable safety and good immunogenicity for healthy Chinese infants. In order to evaluate the efficacy of the vaccine against Hand, Foot and Mouth disease caused by EV71, and to further explore the safety profile of this vaccine in expending infant population, a phase III clinical trial is planed to conduct.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, aged from 6 months to 11 years old Health is determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator
* Provided legal identification for the sake of recruitment
* Subjects and/or parent(s)/legal guardian(s) are able to understand and sign informed consents

Exclusion Criteria:

* History of Hand-foot-mouth Disease
* Subject that has allergic history of vaccine, or allergic to any ingredient of vaccine
* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Congenital malformations or developmental disorders, genetic defects, or severe malnutrition
* Epilepsy, seizures or convulsions history, or family history of mental illness
* Autoimmune disease or immunodeficiency, or parents, brothers and sisters have autoimmune diseases or immunodeficiency
* History of asthma, angioedema, diabetes or malignancy
* History of thyroidectomy or thyroid disease that required medication within the past 12 months
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* Asplenia, functional asplenia or any condition resulting in the absence or removal the spleen
* Acute illness or acute exacerbation of chronic disease within the past 7 days
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
* History of any blood products within 3 months
* Administration of any live attenuated vaccine within 14 days
* Administration of subunit or inactivated vaccines ,e.g., pneumococcal vaccine, or allergy treatment within 7 days
* Axillary temperature > 37.0 centigrade before vaccination
* Abnormal laboratory parameters before vaccination
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10077 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The incidence rate of Hand, Foot and Mouth disease caused by EV71 within one year observation period after the second vaccination | From 28 days after the second vaccination to one year
  to evaluate the efficacy of EV71 vacccine against HFMD caused by EV71

SECONDARY OUTCOMES:
The GMT of anti-EV71 antibodies in serum after second vaccination | 28 days after first vaccination
  to evaluate the GMT of anti-EV71 antibodies in serum 28 days after second vaccination
The GMT of anti-EV71 antibodies in serum 7 and 13 months after second vaccination | 7 and 13 months after second vaccination
  to evaluate the immune persistence of anti-EV71 antibodies in serum
Frequency of systemic and local adverse reactions after the first vaccination | 28 days after the first vaccination
  Frequency of systemic and local adverse reactions in healthy infants following first doses of EV71 vaccine
Frequency of systemic and local adverse reactions after the second vaccination | 28 days after the second vaccination
  Frequency of systemic and local adverse reactions in healthy infants following second doses of EV71 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, BS, Principal Investigator — Jiangsu Center for Diseases Control and Prevention
Locations (3):
- China (3):
  - Ganyu, Lianyungang, Jiangsu
  - Taixing, Taizhou, Jiangsu
  - Sheyang CDC, Yancheng, Jiangsu

REFERENCES:
- [Derived] Zhu F, Xu W, Xia J, Liang Z, Liu Y, Zhang X, Tan X, Wang L, Mao Q, Wu J, Hu Y, Ji T, Song L, Liang Q, Zhang B, Gao Q, Li J, Wang S, Hu Y, Gu S, Zhang J, Yao G, Gu J, Wang X, Zhou Y, Chen C, Zhang M, Cao M, Wang J, Wang H, Wang N. Efficacy, safety, and immunogenicity of an enterovirus 71 vaccine in China. N Engl J Med. 2014 Feb 27;370(9):818-28. doi: 10.1056/NEJMoa1304923. PMID 24571754
- [Derived] Chong P, Hsieh SY, Liu CC, Chou AH, Chang JY, Wu SC, Liu SJ, Chow YH, Su IJ, Klein M. Production of EV71 vaccine candidates. Hum Vaccin Immunother. 2012 Dec 1;8(12):1775-83. doi: 10.4161/hv.21739. Epub 2012 Sep 19. PMID 22992566